CLINICAL TRIAL: NCT00230464
Title: A Double-Blind, Placebo-Controlled, Randomized, Crossover Study to Explore the Acute Effects of LAF 237 on the Rate of Appearance and Disappearance of Glucose During the Overnight Post-Absorptive Period in Type 2 Diabetics
Brief Title: Acute Metabolic Effects of LAF 237 in Type 2 Diabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CLAF237A2346
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2006-01-04 (Estimated); Status verified 2005-09

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; rate of appearance of glucose; insulin secretion; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine

INTERVENTIONS:
Drug: LAF 237

SUMMARY:
Incretin hormones (GIP and GLP-1) stimulate insulin release in a glucose dependant manner, hence are necessary for maintenance of normal glucose tolerance. Both GIP and GLP-1 are degraded and inactivated by DPP-4.

LAF 237 is an inhibitor of DPP-4 that has been shown to increase meal-stimulated levels of intact GLP-1 in animals and patients with T2DM..

The purpose of the current study is to explore the acute effects of LAF237 on the rate of appearance and disappearance of glucose in type 2 diabetics. Secondary objectives include the effect on FPG, insulin secretion rates, glucagon and FFA levels, and rate of glucose entry from the GI tract.

DETAILED DESCRIPTION:
Study Design Double blind, placebo-controlled, randomized, two -period crossover study. Sixteen (16) both sexes diabetic patients will be enrolled and randomized to receive one of two treatment sequences (LAF-placebo or placebo-LAF).

At screening, patients will begin a weight maintaining diet containing 50% carbohydrates, 30% protein and 20% fat.

Within 7 days from screening patients will be scheduled for treatment 1. Patients will begin a 10-hour overnight fast on Day -1 at ~21h00. Patients will be admitted to GCRC next day. Fasting plasma glucose sample will be drawn and following this the patient will be served a standard breakfast containing 1/5 of their caloric allotment (50% carbohydrates, 30% protein and 20% fat). At noon patient will be fed a standard lunch containing 2/5 of their caloric allotment (50% carbohydrates, 30% protein and 20% fat). At 14h30 (-210) an infusion of 3-3H glucose will be started and continued until 08h00 next day (20 µCi x FPG/100 continuous, 0.20/min). At 17h30 (-30) patients will ingest 100 mg of LAF237 or placebo with 200 ml of water. At 18h00 (time zero) patients will be served a dinner (2/5 of their caloric allotment). The carbohydrates (glucose) in the meal will be labeled with 75 µCi of [1-14C]-glucose.

At -60, -50, -40, -35, -30, -20, -10, -5, and 0 minutes before dinner plasma samples for determination of glucose, insulin, C-peptide, glucagons, GLP-1, GIP, FFA, lactate, and amino acid concentrations and 3-3H glucose radioactivity will be drawn. Following dinner, further blood samples will be drawn every 15 minutes for 3.5 hours (18h00-21h30) and every 30 minutes for the next 10.5 hours (22h00-08h00 Day 2). Post dinner samples will be analyzed for the above parameter as well as for 14C glucose radioactivity. At 08h00 on Day 2, both catheters will be removed and the patients will be fed breakfast and then released from the site.

In addition to blood samples, urine from dinner time until 08h00 on Day 2 will be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years with type 2 diabetes, males or females (non-pregnant)
2. Time of diagnosis: within 6 months prior to screening, or 1 month prior to screening with no detectable anti-GAD Abs
3. Normal physical exam, EKG, blood tests, and urinalysis
4. HbA1c=7-11% at screening
5. FPG=160-280 mg/dl at screening
6. Diabetes controlled by diet and exercise alone or by stable dosage of metformin or sulfonylurea
7. BMI=22-45 kg/m2 and with a stable (+/- 2.5 kg) weight for the last 6 months
8. Compliant to study requirements & written consent.

Exclusion Criteria:

1. Pregnant or lactating female
2. History of: type 1 DM, pancreatic injury, secondary diabetes (Cushing, acromegaly), acute metabolic complications (ketoacidosis or hyperosmolar state) within the past 6 months, torsades des pointes, ventricular tachycardia or ventricular fibrillation
3. Any of the following within the past 6 months: MI, CABG, unstable angina
4. ECG abnormalities: second degree AV block (Mobitz 1 and 2), third degree AV block, prolonged QTc (>450 ms)
5. Use of the following medications: class Ia ,Ib, Ic or III antiarrhythmics, insulin, thiazolidinediones, corticosteroids
6. Investigational drug treatment within 4 weeks prior to screening unless local health authority guidelines mandate a longer period
7. Fasting triglycerides >700 mg/dl at screening
8. Diabetic complications
9. Renal disease (creatinine >1.5 mg/dl-males or >1.4 mg/dl-female), renal failure, hepatic dysfunction, thyrotoxicosis
10. History of gastrointestinal surgery (partial bowel resections, partial gastric resections)
11. Donation of one unit of blood within 2 weeks or transfusion within 8 weeks prior to screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16
Dates: Start 2004-11; Study Completion 2005-09

PRIMARY OUTCOMES:
Rate of appearance of endogenous glucose

SECONDARY OUTCOMES:
Rate of dissapearance of glucose
Fasting glucose
Insulin secretion
Free fatty acids
Glucagon
Rate of appearance of oral glucose

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A DeFronzo, MD, Principal Investigator — University of Texas
Locations (1):
- Audie L Murphy VA Hospital, San Antonio, Texas, United States